CLINICAL TRIAL: NCT03712956
Title: CAELYX® as Adjuvant Treatment in Early Stage Luminal B Breast Cancer: a Feasibility Phase II Trial
Brief Title: CAELYX® as Adjuvant Treatment in Early Stage Luminal B Breast Cancer BREAST CANCER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Collaborators: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 0062
Record Dates: First submitted 2018-09-25; First posted 2018-10-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: early breast cancer; luminal B; adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caelyx® for 8 courses (Experimental): Caelyx® administered intravenously at a dose of 20 mg/m2 once every two weeks for 8 courses.
  Interventions: Drug: Caelyx®

INTERVENTIONS:
Drug: Caelyx® — Caelyx® every two weeks for 8 courses
  Other Names: Caelyx

SUMMARY:
A single-center, phase II, single-arm, feasibility study to evaluate PLD (Caelyx®) as an adjuvant chemotherapy regimen in patients with early-stage luminal B breast cancer.

The primary endpoint will be to evaluate the feasibility of adjuvant PLD (Caelyx®) for each individual subject. The regimen will be considered feasible if that subject is able to achieve relative dose intensity (RDI) of at least 85% of the 8 cycles of treatment.

Caelyx® should be administered intravenously at a dose of 20 mg/m2 once every two weeks for 8 courses.

DETAILED DESCRIPTION:
In the 2011 St Gallen Consensus Conference, the Panel considered that both anthracyclines and taxanes should be included in the chemotherapy regimen for 'Luminal B' disease1. However, several patients are reluctant to receive a "strong" chemotherapy because of the fear of its toxic effects, and usually ask for a somehow "less intensive" approach, even accepting a possible reduction in the treatment efficacy.

One of the reasons why patients refuse chemotherapy more often is the fear of alopecia. Few dermatologic conditions carry as much emotional distress as chemotherapy-induced alopecia. Hair loss negatively affects a patient's perception of appearance, body image, sexuality, and self- esteem.

We decided to conduct a single-center, phase II, single-arm, feasibility study to evaluate PLD (Caelyx®) as an adjuvant chemotherapy regimen in patients with early-stage luminal B breast cancer.

The primary endpoint will be to evaluate the feasibility of adjuvant PLD (Caelyx®) for each individual subject. The regimen will be considered feasible if that subject is able to achieve relative dose intensity (RDI) of at least 85% of the 8 cycles of treatment.

Secondary endpoints will include:

* Adverse events
* Tolerability (treatment completion)
* Breast cancer free interval (BCFI; events are reappearance of invasive breast cancer at any site including contralateral disease)
* Disease Free Survival (DFS) (includes second malignancies and deaths)
* Overall survival (OS) Caelyx® should be administered intravenously at a dose of 20 mg/m2 once every two weeks for 8 courses.

ELIGIBILITY:
Inclusion Criteria:

* Performance status (ECOG) 0-2
* Operable histologically confirmed breast cancer
* Luminal B HER2-negative (ER positive, HER2 negative, and at least one of the following:

Ki- 67 'high' (≥20%) or PgR 'negative or low') or Luminal B HER2-positive (ER positive, HER2 over-expressed or amplified, any Ki-67, any PgR)

* Early-stage (pT1-3; any nodal status)
* Candidate to adjuvant chemotherapy and endocrine therapy
* The tumor must be confined to the breast and axillary nodes without detected metastases elsewhere
* Patients with synchronous (diagnosed histologically within 2 months) bilateral invasive breast cancer are eligible if all other criteria are met
* Patients must have had surgery for primary breast cancer with no known clinical residual loco-regional disease
* Margins must be negative for invasive breast cancer and DCIS
* Patients should start treatment as close to definitive surgery as possible (no later than 8 weeks)
* No prior neoadjuvant or adjuvant therapy for breast cancer. Note: Radiotherapy is allowed prior to trial entry. Raloxifene, tamoxifen, or other SERM must be discontinued at least 4 weeks before trial entry.
* No hormone replacement therapy (HRT)
* No hormonal therapy, except steroids for adrenal failure, hormones for non-breast cancer related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic.
* No treatment with bisphosphonates, except for the treatment of osteoporosis
* Adequate bone marrow, renal, and hepatic function must be assessed within 2 months before trial entry and values must meet the following criteria:
* WBC ≥ 3.0 x 109/L
* Granulocyte count ≥ 1.500 x 109/L
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥ 100 x 109/L
* Serum creatinine < 1.35 mg/dl - Calculated creatinine clearance at least 50 mL/min
* Serum bilirubin within normal/reference range
* AST/ALT within 1.5 x upper normal limit

  * Adequate cardiovascular function defined as the following must be assessed within 2 months before trial entry:
* LVEF ≥ 50% by echocardiography, radionuclide ventriculography or Multigated Angiography (MUGA) - No ECG evidence of acute ischemia
* No evidence of medically relevant conduction system abnormalities, which in the opinion of the investigator would preclude trial entry
* No myocardial infarction within the past 6 months
* No New York Heart Association (NYHA) class III or IV congestive heart failure
* Negative pregnancy test (in fertile women).
* Written Informed Consent (IC) must be signed and dated by the patient and the investigator prior to trial entry.
* Patients must be accessible for follow-up.
* Patients should have no psychiatric, addictive, or cognitive disorder that would prevent compliance with protocol requirements.

Exclusion Criteria:

* Patients with a history of any prior ipsilateral or contralateral invasive breast cancer.
* Patients with previous or concomitant malignancy diagnosed within the past five years. Patients with adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, contra- or ipsilateral in situ breast carcinoma are eligible regardless of the date of diagnosis.
* Patients with other non-malignant uncontrolled systemic diseases that would preclude trial entry in the opinion of the investigator. Specifically not eligible are patients with uncontrolled active infection, chronic infection such as active HBV or HCV.
* Patients with myocardial infarction or pulmonary embolism within 6 months prior to trial entry.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2016-03-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of adjuvant PLD (Caelyx®) | 4 months
  The regimen will be considered feasible if that subject is able to achieve relative dose intensity (RDI) of at least 85% of the 8 cycles of treatment

SECONDARY OUTCOMES:
Adverse event | 4 months
  Grading for all side effects will be according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
percent of patient completing treatment (tolerability) | 4 month
  percent of patients treated according to the protocol and completing the adjuvant program, and percent protocol treatment received
Breast cancer free interval (BCFI) | 5 years
  BCFI is defined as the time from registration to local (including recurrence restricted to the breast after breast conserving treatment), regional, or distant relapse, or contralateral breast cancer.
Disease Free Survival (DFS) | 5 years
  DFS is defined as the time from registration to disease recurrence (includes second malignancies and deaths)
Overall survival (OS) | 5 years
  OS defined as the time from registration to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Munzone, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No